CLINICAL TRIAL: NCT01571726
Title: Novel Imaging Modalities to Characterize Angiogenesis in the Bone Marrow Microenvironment in Multiple Myeloma (MM) and Its Precursor Disease
Brief Title: Imaging Studies and the Development of Multiple Myeloma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 120106; 12-C-0106
Record Dates: First submitted 2012-04-04; First posted 2012-04-05 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2014-04-16

CONDITIONS: Multiple Myeloma; Smoldering Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance
Keywords: (18)-Fluciclatide PET/CT; Serum M-Protein; Percentage of Plasma Cells in the Bone Marrow; Ratio of Normal/Abnormal Percentage of Plasma Cells in the Bone Marrow; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Smoldering Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance | interventions — AH 111585

INTERVENTIONS:
Drug: Fluciclatide — 7mCi

SUMMARY:
Background:

- Multiple myeloma (MM) is a type of malignant blood cancer. It affects the plasma cells, which help produce antibodies and fight infection. MM is nearly always preceded by a pre-malignant state, monoclonal gammopathy of undetermined significance (MGUS) or smoldering multiple myeloma (SMM). Currently, it is not possible to predict when someone with MGUS or SMM will develop MM. Also, the disease changes in those early states are not well understood. Researchers want to look at imaging studies of people with MGUS, SMM, and MM. They will study whether the growth of blood vessels can be used to predict disease progression.

Objectives:

- To use imaging studies to evaluate disease progression in multiple myeloma.

Eligibility:

- Individuals at least 18 years of age who have MGUS, SMM, or newly diagnosed MM.

Design:

* Participants will be screened with a physical exam and medical history. They will also have blood and urine tests, and provide bone marrow samples.
* Participants will have positron emission tomography (PET) scans with the new contrast agent [18]F-Fluciclatide. The contrast agent is intended to show patterns of increased vessel growth in the bone marrow.
* Participants will also have a magnetic resonance imaging (MRI) scan. This scan will be done according to standard procedures.
* Researchers will compare these scans with blood tests and other clinical information to study disease progression of MGUS, SMM, and MM.

DETAILED DESCRIPTION:
Background:

* Multiple myeloma (MM) is a plasma cell neoplasm with a median survival of 3-4 years.
* Monoclonal gammopathy of undetermined significance (MGUS) and smoldering myeloma (SMM) are premalignant plasma cell proliferative disorders characterized by elevated monoclonal protein and bone marrow plasma cells. MGUS affects 3.2% of Caucasians over the age of 50 and has a 1% annual risk of progression to MM. Approximately 3,000 cases of SMM are diagnosed annually with a 10% annual risk of progression to MM.
* Currently, it is not possible to predict which patients will progress to MM, and the biological changes occurring in those precursor states remain poorly understood.
* Angiogenesis is a hallmark of multiple myeloma and its precursor disease.

Angiogenesis has been measured using microvessel density. In a prior study, we have demonstrated increased microvessel density using CD34 immunohistochemistry in patients with multiple myeloma, compared to SMM or MGUS, suggesting that there is increased vascular density as the disease progresses. A correlation between MM disease stage and prognosis has been reported for several serum angiogenic factors and myeloma cells and bone marrow endothelial cells have been shown to secrete and respond to angiogenic modulators.

* Dynamic contrast-enhanced (DCE)-MRI is a noninvasive way to evaluate angiogenesis. In a prior NIH study, we have demonstrated that the kep (a measure of contrast influx in vessels in the bone marrow microenvironment) to be gradually higher in MM>SMM>MGUS, however it was limited to imaging a single field of view (i.e. the lumbar spine). This is also highly correlated with microvessel density.
* Fluciclatide is a small cyclic peptide containing the RGD tri-peptide, which preferentially binds with high affinity to Alpha(v)Beta(3) integrins, which are up-regulated in angiogenesis.
* Alpha(v)Beta(3) integrins are also expressed on certain types of tumor cells and on activiated osteoclasts.
* (18)Fluciclatide (previously known (18)F-AH111585) is a new radiopharmaceutical developed for PET imaging, which targets Alpha(v)Beta(3) receptors.
* Novel imaging modalities using tracers specific for angiogenesis, using (18)F-Fluciclatide whole-body PET/CT imaging may improve our ability to predict patients who are at high risk of progression.

Objectives:

* The primary objective of the study is to explore the distribution of (18)F-Fluciclatide PET/CT in bone marrow microenvironment in patients with multiple myeloma and its precursor disease.
* The secondary objectives are to preliminarily evaluate the distribution of (18)Fluciclatide PET/CT with respect to DCE-MRI and bone marrow vascularity determined by immunohistochemistry (CD34) on the bone marrow biopsy specimen.
* To preliminarily evaluate the distribution of (18)F-Fluciclatide PET/CT with respect to established clinical markers of progression from MGUS/SMM to MM, including serum M-protein, percentage of plasma cells in the bone marrow, serum free light-chain abnormalities and immunoparesis, and ratio of normal/abnormal plasma cells in the bone marrow by flow cytometry.

Eligibility:

* A confirmed diagnosis of MGUS, SMM or MM (based on IMWG diagnostic criteria)
* Age greater than or equal to 18 years
* ECOG performance status in the range of 0-2

Design:

* This is a cross-sectional pilot study of patients with MGUS, SMM or MM.
* Subjects with frank multiple myeloma will be enrolled first. If the (18)F-Fluciclatide PET/CT is negative in the first 5 subjects, the study will be aborted and we will not proceed with MGUS or SMM patients. However if the 18F-Fluciclatide PET/CT is positive in MM patients, then we will proceed with MGUS and SMM patients.
* Subsequently (18)F-Fluciclatide PET/CT and DCE-MRI imaging will be done in all the patients. When feasible, an optional non-contrast wholebody MR may also be performed.
* 10 MM, 10 SMM and 10 MGUS patients will be enrolled on this protocol.
* Patients may donate cellular products or tissues as appropriate for research purposes.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Diagnosis of MGUS, SMM and MM will be made in accordance with the clinical diagnostic criteria set forth by the International Myeloma Working Group. The diagnosis will be confirmed by the following diagnostic tests:

  * serum/urine protein electrophoresis
  * serum/urine immunofixation,
  * light-chain assays,
  * a skeletal survey, or
* immunohistochemistry analyses of the bone marrow biopsy, or
* a combination of these at the NIH

Note: Written results from institutions outside of NIH for the above tests will be accepted if available.

* Age greater than or equal to 18 years.
* ECOG performance status of 0-2.
* The patient must be competent to sign an informed consent form.
* Platelet count = or > 100,000. Subjects must weight <320lbs
* Creatinine <2.5 times ULN or eGFR>30 ml/min/1.73m(2)

EXCLUSION CRITERIA:

* A medical history of other malignancy (apart from basal cell carcinoma of the skin or in situ cervical carcinoma; also, for MM patients this does not include MM) except if the patient has been free of symptoms and without active therapy during at least the previous 3 years.
* Patients with documented metastatic lesions from another type of malignancy will be excluded.
* Female subject is pregnant or breast-feeding.
* The subject has known allergy to gadolinium
* The subject has contraindications to MRI

  * Subjects must weigh <136 kg (weight limit for scanner table).
  * Subjects cannot have pacemakers, cerebral aneurysm clips, shrapnel injury, or other implanted electronic devices or metal not compatible with MRI.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03-27; Primary Completion 2014-04-23 (Actual); Study Completion 2014-04-23 (Actual)

PRIMARY OUTCOMES:
To explore the distribution of 18F-Fluciclatide PET/CT in bone marrow microenvironment in patients with multiple myeloma and its precursor disease (MGUS and SMM) | 1 year

SECONDARY OUTCOMES:
Distribution of agent | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Carl O Landgren, M.D., Principal Investigator — National Cancer Institute (NCI)

REFERENCES:
- [Background] Kyle RA, Rajkumar SV. Multiple myeloma. Blood. 2008 Mar 15;111(6):2962-72. doi: 10.1182/blood-2007-10-078022. PMID 18332230
- [Background] International Myeloma Working Group. Criteria for the classification of monoclonal gammopathies, multiple myeloma and related disorders: a report of the International Myeloma Working Group. Br J Haematol. 2003 Jun;121(5):749-57. PMID 12780789
- [Background] Kumar SK, Rajkumar SV, Dispenzieri A, Lacy MQ, Hayman SR, Buadi FK, Zeldenrust SR, Dingli D, Russell SJ, Lust JA, Greipp PR, Kyle RA, Gertz MA. Improved survival in multiple myeloma and the impact of novel therapies. Blood. 2008 Mar 1;111(5):2516-20. doi: 10.1182/blood-2007-10-116129. Epub 2007 Nov 1. PMID 17975015